CLINICAL TRIAL: NCT00663416
Title: A Phase IIb Prospective, Randomized, Double-blind, Placebo Controlled Study of NTx™-265: Human Chorionic Gonadotropin (hCG) and Epoetin Alfa (EPO) in Acute Ischemic Stroke Patients (REGENESIS)
Brief Title: REGENESIS (CA): A Study of NTx™-265: Human Chorionic Gonadotropin (hCG) and Epoetin Alfa (EPO) in Acute Ischemic Stroke Patients
Acronym: REGENESIS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Stem Cell Therapeutics Corp. (Industry)
Responsible Party: Alan Moore / President & Chief Executive Officer, Stem Cell Therapeutics Corp.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NTx™-265-CP-201-IS (CA)
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Last update posted 2009-08-12 (Estimated); Status verified 2009-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Ovidrel; Epoetin Alfa; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: NTx™-265: rhCG, then rEPO
- 2 (Placebo Comparator)
  Interventions: Drug: Saline placebo

INTERVENTIONS:
Drug: NTx™-265: rhCG, then rEPO — * rhCG 10,000 IU, SC, on Day 1, 3, and 5 of study participation, then
  * rEPO 30,000 IU, IV, on Day 7, 8, and 9 of study participation
  Other Names: Ovidrel; Eprex
  Arms: 1
Drug: Saline placebo — * Saline SC, on Day 1, 3, and 5 of study participation, then
  * Saline IV, on Day 7, 8, and 9 of study participation
  Other Names: Sodium Chloride 0.9%
  Arms: 2

SUMMARY:
Primary objective: To assess the neurological outcome in acute ischemic stroke patients treated with NTx™-265, when compared with patients given a placebo control.

Secondary objective: To assess the safety and tolerability of NTx™-265 when given to acute ischemic stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85.
* NIHSS score 6-24 within 24-48 hours after stroke onset and enrolment.
* Stroke is ischemic in origin, supratentorial, and radiologically confirmed (CT scan or diagnostic MRI) prior to enrolment.
* Patient is 24-48 hours from time of stroke onset when the first dose of NTxTM-265 therapy is administered. Time of onset is when symptoms began; for stroke that occurred during sleep, time of onset is when patient was last seen or was self-reported to be normal.
* Reasonable expectation of availability to receive the full 9 day NTxTM-265 course of therapy, and to be available for subsequent follow-up visits.
* Reasonable expectation that patient will receive standard post-stroke physical, occupational and speech therapy as indicated.
* Female patient is either:

  1. Not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile (bilateral oophorectomy or hysterectomy) or
  2. If of childbearing potential, agrees to use two of the following effective separate forms of contraception throughout the study, up to and including the follow-up visits:

     * Condoms, sponge, foams, jellies, diaphragm or intrauterine device, contraceptives (e.g., implants, injectables, combined oral, etc) OR
     * A vasectomised partner OR
     * Abstinence

Exclusion Criteria

* Patients presenting with lacunar, hemorrhagic and/or brain stem stroke.
* Patients who have received thrombolytic treatment with tPA following the index stroke.
* Patients classified as comatose, defined as a patient who required repeated stimulation to attend, or is obtunded and requires strong or painful stimulation to make movements (NIHSS 1A score must be <2)
* Women who have tested positive for pregnancy, or are breast-feeding or are not using a highly effective method of birth control that can be maintained for the duration of the study.
* Serum hemoglobin > 16 g/dL (males) or > 14 g/dL (females); or platelet count > 400,000/mm3.
* Advanced liver,kidney, cardiac or pulmonary disease; the former will be operationally defined using NCI Toxicity Criteria (Grade 2 or higher)
* Serum bilirubin > 1.5 x upper limit of normal (ULN).
* Alkaline phosphatase > 2.5 x ULN.
* AST>2.5xULN.
* ALT > 2.5 x ULN.
* Creatinine > 2.0 x ULN.
* Patients with known and documented transferrin saturation < 20%.
* Patients with known and documented ferritin < 100 ng/mL.
* Patients with known and documented elevated PSA levels, or a PSA level of ≥ 4 ng/mL at screening.
* Patients with a known or current history of abnormal hypercoagulability parameters , including known cardiolipin/antiphospholipid antibody syndrome.
* Expected survival < 1 year.
* Allergy or other contraindication to hCG including:

  1. Prior hypersensitivity to hCG preparations or one of their excipients.
  2. Primary ovarian failure.
  3. Uncontrolled thyroid or adrenal dysfunction.
  4. An uncontrolled organic intracranial lesion such as a pituitary tumor.
  5. Abnormal uterine bleeding of undetermined origin.
  6. Ovarian cyst or ovarian enlargement of undetermined origin.
  7. Sex hormone dependent tumors of the reproductive organs, accessory sex glands, and breasts.
* Allergy or other contraindication to epoetin alfa:

  1. Who developed pure red cell aplasia following treatment with any erythropoiesis regulating hormones
  2. With uncontrolled hypertension
  3. With known hypersensitivity to mammalian cell-derived products, albumin (human) or any component of the product
  4. Who for any reason cannot receive adequate antithrombotic treatment
* A known diagnosis of cancer (except non-malignant skin cancer).
* Uncontrolled hypertension, defined in the context of acute stroke as blood pressure persistently above 220 mm Hg systolic or 120 mm Hg diastolic despite antihypertensive therapy.
* Use of either hCG or epoetin alfa within the previous 90 days.
* Any condition known to elevate hCG, active in the prior 24 months, e.g., choriocarcinoma or germ cell tumor.
* Patients with a pre-stroke/pre-morbid modified Rankin Score (mRS) ≥ 2.
* Any patients living in a nursing home or supervised living center. Patients must be historically fully independent in all activities of daily living including banking, shopping, cooking, toileting, showering and dressing.
* Any other medical condition or degree of stroke such that, in the investigator's opinion, the patient should not be included in the trial.
* With the exception of the qualifying stroke, any other stroke within the previous 6 months.
* Patients who cannot take anti-platelet therapy for the duration of the study.
* Patients who cannot take low molecular weight or unfractionated heparin during hospitalization.
* Pre-existing and active major psychiatric or other chronic neurological disease.
* Consume, on average, greater than 14 alcoholic drinks per week, or have a history of substance abuse or dependency within 12 months prior to the study.
* Currently participating in another investigational study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-10 (Estimated); Study Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Score (mRS) | Day 90
NIHSS response | Day 90

SECONDARY OUTCOMES:
NIHSS | Day 90
mRS | Day 90
Barthel Index | Day 90
Action Research Arm Test | Day 90
Gait Velocity Test | Day 90
Boston Naming Test | Day 90
Line Cancellation Test | Day 90
Trails A & B Test | Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Hill, MD, Principal Investigator — Department of Clinical Neurosciences, University of Calgary; Steven C Cramer, MD, Principal Investigator — Department of Neurology, University of Califonia, Irvine Medical Center
Locations (26):
- Canada (16):
  - Department of Clinical Neurosciences, Univeristy of Calgary, Calgary, Alberta
  - Walter Mackenzie Health Sciences Centre, Edmonton, Alberta
  - Grey Nuns Community Hospital, Edmonton, Alberta
  - Chinook Regional Hospital, Lethbridge, Alberta
  - Penticton Regional Hospital, Penticton, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Vancouver Island Health Research Centre, Victoria, British Columbia
  - Brandon Regional Health Centre, Brandon, Manitoba
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - McMaster Clinic, Hamilton, Ontario
  - Trillium Health Centre, Mississauga, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Division of Neurology , Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Department of Neurology, St. Michael's Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Montreal Neurological Institute, Montreal, Quebec
- India (10):
  - Department of Neurology, Care Hospital, Hyderabad, Andhra Pradesh
  - Krishna Institute of Medical Sciences, Hyderabad, Andhra Pradesh
  - Department of Neurology, Apollo Hospitals, Hyderabad, Andhra Pradesh
  - Department of Neurology, Nizam's Institute of Medical Science, Hyderabad, Andhra Pradesh
  - M S Ramaiah Memorial Hospital, Bangalore, Karnataka
  - Max Super Speciality Hospital, New Delhi, National Capital Territory of Delhi
  - Christian Medical College & Hospital, Ludhiana, Punjab
  - Department of Neurology, Christian Medical College, Vellore, Tamil Nadu
  - AMRI Hospital, Kolkata, West Bengal
  - Department of Neurology, B.P.Poddar Hospital & Medical Research Ltd, Kolkata, West Bengal